CLINICAL TRIAL: NCT04702243
Title: Defining the Genetic Etiology of Suppurative Lung Disease in Children and Adults
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Washington University School of Medicine (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Children's Hospital Colorado (Other); Stanford University (Other); Seattle Children's Hospital (Other); The Hospital for Sick Children (Other); McGill University (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 20-0508; 5U54HL096458-17 (NIH)
Record Dates: First submitted 2020-12-16; First posted 2021-01-08 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Primary Ciliary Dyskinesia; Primary Immune Deficiency; Kartagener Syndrome
MeSH Terms: conditions — Ciliary Motility Disorders; Primary Immunodeficiency Diseases; Kartagener Syndrome | interventions — Genetic Testing; Apoptosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood draw or buccal swab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Affected Participants: Subjects who have suppurative lung disease without a known genetic diagnosis
  Interventions: Diagnostic Test: Genetic Testing for PCD or PID
- Unaffected Family Members: Unaffected family members may be enrolled in the study for collection of DNA only
  Interventions: Other: Unaffected Family Member Genetic Testing

INTERVENTIONS:
Diagnostic Test: Genetic Testing for PCD or PID — Patients with high likelihood of a PID disorder or a high likelihood of PCD will initially undergo research genetic testing on a commercial approved panel for PID disorders or a panel of at least 37 PCD genes.
  Groups: Affected Participants
Other: Unaffected Family Member Genetic Testing — Unaffected family members will undergo genetic testing if genetic findings are identified in their affected family member.
  Groups: Unaffected Family Members

SUMMARY:
The investigators will utilize a systematic approach for the diagnostic evaluation of patients to identify characteristics which may distinguish between Primary Immunodeficiency (PID) disorders versus Primary Ciliary Dyskinesia (PCD).

DETAILED DESCRIPTION:
This protocol utilizes a cross-sectional study design. Over a 5-year period, the investigators will enroll patients who have clinical and lab features characteristic of a PID disorder or PCD, but do not have a confirmed genetic diagnosis. Innovative, standardized methods (SOPs) will be utilized, including ciliary ultrastructural analyses by transmission electron microscopy (TEM), as pertinent. Measures of nasal nitric oxide (nNO) will be performed in all subjects to allow comparisons of nNO values in PID vs. PCD. Patients with high likelihood of a PID disorder or a high likelihood of PCD will initially undergo research genetic testing on a commercial approved panel for PID disorders or a panel of at least 37 PCD genes. All subjects who do not have a genetic diagnosis from the test panels will undergo whole exome sequencing (WES) to search for novel genetic etiologies for PID or PCD.

ELIGIBILITY:
Pediatric subjects (aged 5-17 years): Inclusion criteria include the major criterion (bronchiectasis in > 1 lobe on current or chest CT in previous 24 months, if available for review), plus one minor criterion, or two minor criteria, if bronchiectasis is not present, (including at least 1 "lung" minor criteria).

Adult subjects (aged 18-45 years): Inclusion criteria include the major criteria (bronchiectasis in > 1 lobe on current or chest CT in previous 36 months, if available for review), plus one minor criterion, or three minor criteria, if bronchiectasis is not present, (including at least 1 "lung" minor criteria).

Inclusion Criteria:

General Criteria

* Age 5-45 years
* Male and Female Subjects
* All races and ethnicities

Major Clinical Criteria

- Bronchiectasis in > 1 lobe

Minor Clinical Criteria, Lung

* Neonatal respiratory distress (in term neonates with O2 requirement)
* Chronic wet cough (year-round for at least 12 months)
* Recurrent episodes of bacterial bronchitis
* Recurrent pneumonia (confirmed on chest x-ray)
* Respiratory non-tuberculous mycobacteria (NTM) (documented respiratory NTM culture)

Minor Clinical Criteria, Other

* Chronic nasal congestion
* Recurrent/chronic paranasal sinusitis
* Ongoing middle-ear disease and/or tympanostomy tube placement at age ≥ 4 years
* Organ laterality defect
* Low nasal nitric oxide (< 77 nL/min) (by plateau measurement)
* Confirmed family history of PID or PCD

Exclusion Criteria:

* Anyone who has a confirmed genetic diagnosis of PCD or PID
* Cystic Fibrosis
* Alpha-antitrypsin deficiency in adults (18 years and older)
* Congenital upper or lower airway anomalies
* Post-lung or heart transplant, or other conditions requiring immunosuppression therapy
* Other confounding features, such as lung disease due to prematurity (born < 28 weeks gestation) or HIV
* Neurological compromise and evidence of recurrent aspiration
* Conditions known to be commonly associated with bronchiectasis, such as prior mycobacterium tuberculosis
* Have not had standard clinical evaluation to address other potential causes of chronic oto-sino- pulmonary disease, particularly cystic fibrosis, aspiration or airway anatomic abnormalities.

Ages: 5 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects who have suppurative lung disease but without a defined genetic diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 436 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-08-06 (Actual); Study Completion 2025-08-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants with a Confirmed Diagnosis of PCD or PID | Up to approximately 4 years
  A commercial genetic panel will be used to test for disease causing mutation in PCD or PID. If the commercial panel does not yield positive results, WES research testing will be used to identify disease causing mutations in PCD and PID in order to confirm the diagnosis.
Prevalence of Neonatal Respiratory Distress Seen in PCD and PID | During a single 6-hour visit
  Medical records will be reviewed to denote presence or absence of neonatal respiratory distress (occurs at birth).
Prevalence of the Onset of Chronic Nasal Congestion Before Six Months of Age Seen in PCD and PID | During a single 6-hour visit
  Medical records will be reviewed to denote presence or absence of the onset of chronic nasal congestion before age 6 months.
Prevalence of the Onset of Daily Wet Cough Before Six Months of Age Seen in PCD and PID | During a single 6-hour visit
  Medical records will be reviewed to denote presence or absence of the onset of daily wet cough before age 6 months.
Prevalence of Laterality Defects Seen in PCD and PID | During a single 6-hour visit
  Medical records will be reviewed to denote presence or absence of laterality defects (situs inversus/heterotaxy).
Prevalence of Chronic/Recurrent Sinus Disease Seen in PCD and PID | During a single 6-hour visit
  Medical records will be reviewed to denote presence or absence of chronic/recurrent sinus disease.
Prevalence of Chronic/Recurrent Middle Ear Disease Seen in PCD and PID | During a single 6-hour visit
  Medical records will be reviewed to denote presence or absence of chronic/recurrent middle ear disease.
Prevalence of Recurrent Pneumonia/Sepsis Seen in PCD and PID | During a single 6-hour visit
  Medical records will be reviewed to denote to denote presence or absence of recurrent pneumonia/sepsis (that is not bronchiectasis).
Prevalence of Skin Infections/Abscesses Seen in PCD and PID | During a single 6-hour visit
  Medical records will be reviewed to denote to denote presence or absence of skin infections/abscesses.
Prevalence of Abnormal Nasal Nitric Oxide Values Seen in PCD and PID | During a single 6-hour visit
  Nasal nitric oxide will be measured to determine the number of subjects who have an abnormal value, utilizing a cut-off of 77 nl/min.
Prevalence of Abnormal Immunoglobulin G Values Seen in PCD and PID | During a single 6-hour visit
  Immunoglobulin G will be measured to determine the number of subjects who have an abnormal value, utilizing the local laboratory age-defined cut-off ranges (United States: mg/dL; Canada: g/L).
Prevalence of Abnormal Lymphocyte Markers Seen in PCD and PID (Laboratory Tests) | During a single 6-hour visit
  Lymphocyte Markers will be measured to determine the number of subjects who have an abnormal value, utilizing the local laboratory age-defined cut-off ranges (% of lymphocytes).
Mean FEV1 Percent Predicted Values in PCD and PID | During a single 6-hour visit
  Forced expired volume in 1 second (FEV1) will be assessed by percentage of the predicted value (0-100%).

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Olivier, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (8):
- United States (6):
  - Stanford University, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - National Heart, Lung and Blood Institute, Bethesda, Maryland
  - Washington University in St. Louis, St Louis, Missouri
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Seattle Children's Hospital, Seattle, Washington
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - McGill University, Montreal, Quebec